CLINICAL TRIAL: NCT05600868
Title: The Effect of Dual Attention in an EMDR Intervention for Posttraumatic Symptomatology: a Randomized Clinical Trial
Brief Title: The Effect of Dual Attention in an EMDR Intervention
Acronym: DA_EMDR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUP
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Trauma, Psychological; Traumatic Stress Disorder
Keywords: Trauma; Traumatic Stress Disorder; EMDR; Dual Attention
MeSH Terms: conditions — Psychological Trauma; Stress Disorders, Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EMDR+dual attention (Active Comparator): .Processing the trauma with exposition and dual attention.
  Interventions: Behavioral: A comprehensive third-generation intervention EMDR + dual attention
- EMDR + fixed point (Active Comparator): Processing the trauma with exposition and fixed point.
  Interventions: Behavioral: A comprehensive third-generation intervention EMDR + fixed point
- EMDR + exposition (Active Comparator): Processing the trauma with exposition.
  Interventions: Behavioral: A comprehensive third-generation intervention EMDR + dual attention; Behavioral: A comprehensive third-generation intervention EMDR + exposition

INTERVENTIONS:
Behavioral: A comprehensive third-generation intervention EMDR + dual attention — This is a individual intervention with a total of 10 sessions. In the processing the traumatic event phase will be realized with double attention.
  Arms: EMDR + exposition; EMDR+dual attention
Behavioral: A comprehensive third-generation intervention EMDR + fixed point — This is a individual intervention with a total of 10 sessions. In the processing the traumatic event phase will be realized with fixed point.
  Arms: EMDR + fixed point
Behavioral: A comprehensive third-generation intervention EMDR + exposition — This is a individual intervention with a total of 10 sessions. In the processing the traumatic event phase will be realized with exposition.
  Arms: EMDR + exposition

SUMMARY:
Research to date indicates that trauma-focused treatments are safe and effective for PTSD, even when higher-risk comorbidities (e.g., psychosis or substance use) are present. In particular, there are data pointing to the efficacy of prolonged exposure therapy and eye movement desensitization and reprocessing (EMDR) therapy. Clinical practice guidelines specifically recommend trauma-focused treatment with exposure and/or cognitive restructuring components. Regarding EMDR interventions, there are increasing results supporting its efficacy. Some interesting clinical advantages presented by EMDR as opposed to cognitive-behavioral therapies are 1) the efficacy found despite less exposure to the traumatic memory, 2) the exclusion of homework, 3) as well as the rapid reduction in subjective disturbance produced even after a single session of EMDR therapy. However, the mechanisms producing the improvement and, in particular, the effect of bilateral stimulation are not precisely known. More research is needed in this regard since bilateral stimulation is the most controversial part and with less evidence found. In addition to this, there are very few studies that have analyzed the differential efficacy of the presence or absence of bilateral stimulation or of the different types of stimulation possible. As for the comparison between types of stimulation (bilateral with eye movements, or focusing on a fixed point), greater treatment effects have been found for EMDR with fixation on an immobile hand compared to eye movements. The aim of this study is to examine the effectiveness of a comprehensive intervention protocol for people who have experienced traumatic events and present post-traumatic symptomatology. In addition, this study will compare the efficacy of traumatic memory processing with and without dual attention.

DETAILED DESCRIPTION:
The protocol will be developed following the three stages of recovery from trauma: first, focusing on establishing the therapeutic alliance and safety; second, focusing on recounting and re-processing the traumatic event; and third, focusing on reconnecting with others and with life despite the trauma experienced. This study will analyze the differences of type of traumatic processing; 1. using bilateral stimulation, 2. using fixed-point focusing and 3. closing the eyes (only exposure to the traumatic memory, without dual attention).

ELIGIBILITY:
Inclusion Criteria:

* Those showing a high risk of PTSD (TSQ ≥6 or TSQ ≥4 with clinical criteria) will be further evaluated to determine whether they meet the inclusion criteria. Participants must:

  1. Be between the ages of 18 and 65 fluent enough in Spanish language; 2.

Exclusion Criteria:

* Present severe active suicidal ideation, or have made a self-injurious attempt during the last month.
* Present a diagnosis of substance dependence, intellectual disability or severe cognitive dysfunction.
* Participants with a score greater than or equal to 26 on the BDI-II, the inclusion of the person in the study will be assessed by clinical criteria.
* Having received EMDR treatment in the last 6 months.
* Also excluded from the program are those people who cannot guarantee continuity in the therapeutic process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from posttraumatic symptoms at 10 weeks and 6 months | Change baseline, 10 weeks, and 6 months
  International Trauma Questionnaire (ITQ; Cloitre et al., 2018). Higher scores mean a worse outcome.
Change from psychopathological symptoms at 10 weeks and 6 months | Change baseline, 10 weeks, and 6 months
  Symptom Checklist 45-SCL-90R brief (Davison et al., 1997).Higher scores mean a worse outcome.
Change from Dissociative symptoms at 10 weeks and 6 months | Change baseline, 10 weeks, and 6 months
  Dissociative Experience Scale DES II (Carlson and Putnam, 1993). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change from Well-being at 10 weeks and 6 months | Change baseline, 10 weeks, and 6 months
  Scales of Psychological Well-Being (SPWB; Ryff & Keyes, 1995). Higher scores mean a better outcome.
Change from Satisfaction with life at 10 weeks and 6 months | Change baseline, 10 weeks, and 6 months
  Satisfaction with Life Scale (SWLS; Diener et al., 1985).Higher scores mean a better outcome.
Change from Emotion Regulation at 10 weeks and 6 months | Change baseline, 10 weeks, and 6 months
  Cognitive Emotion Regulation Questionnaire (CERQ; Garnefski & Kraaij, 2007).Higher scores mean better outcome for functional dimensions and worse outcome for disfunctional dimensions
Change from Attachment style at 10 weeks and 6 months | Change baseline, 10 weeks, and 6 months
  Psychosis Attachment Measure (PAM; Berry, 2006). Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Carmen Valiente, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code